CLINICAL TRIAL: NCT00376974
Title: The Effect of Patient Education on Glaucoma Medication Compliance
Brief Title: The Effect of Education on Patient Compliance
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: 2006-1
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2006-09-15 (Estimated); Status verified 2006-09

CONDITIONS: Glaucoma
Keywords: glaucoma; compliance; intraocular pressure; video
MeSH Terms: conditions — Glaucoma; Patient Compliance

INTERVENTIONS:
Behavioral: American Academy of Ophthalmology Glaucoma Educational Tape

SUMMARY:
With patient education, the compliance with glaucoma medications will increase.

DETAILED DESCRIPTION:
We divided glaucoma patients into two groups; one watched a video the others did not. We checked their intraocular pressures before and after the intervention to see if there was a difference

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma patients coming in for routine examination

Exclusion Criteria:

* If glaucoma was unstable and treatment regimen required a change

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-03; Study Completion 2006-05

PRIMARY OUTCOMES:
Intraocular pressure

SECONDARY OUTCOMES:
Score on glaucoma educational test

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Orengo-Nania, m.d., Principal Investigator — Baylor College of Medicine
Locations (1):
- MDVAMC, Houston, Texas, United States